CLINICAL TRIAL: NCT02310165
Title: Z-tract Versus Coaxial Insertion Technique in Large Volume Paracentesis
Brief Title: Insertion Technique in Large Volume Paracentesis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Virginia (Other)
Responsible Party: Principal Investigator, Amy Rubin, MD, Department of Gastroenterology, University of Virginia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 16842
Record Dates: First submitted 2014-12-03; First posted 2014-12-05 (Estimated); Last update posted 2014-12-05 (Estimated); Status verified 2014-12

CONDITIONS: Cirrhosis
Keywords: Paracentesis; Ascites
MeSH Terms: conditions — Fibrosis; Ascites

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Z-tract Insertion Technique (Other): For this technique, the skin is pulled 2 cm downward before the paracentesis needle is inserted and advanced.
  Interventions: Procedure: Z-tract Insertion Technique
- Coaxial Insertion Technique (Other): For this technique, the needle is directly inserted to minimize the distance between he cutaneous tissue and ascites
  Interventions: Procedure: Coaxial Insertion Technique

INTERVENTIONS:
Procedure: Z-tract Insertion Technique
  Arms: Z-tract Insertion Technique
Procedure: Coaxial Insertion Technique
  Arms: Coaxial Insertion Technique

SUMMARY:
The purpose of this study is to compare two different methods that are used for inserting the needle during paracentesis. One method is called the "coaxial insertion technique" and the other is called the "z-tract technique". Researchers would like to see which method is better and leads to less problems like oozing from the needle insertion site and pain during the procedure. Both methods are approved and currently used methods for doing a paracentesis at the University of Virginia. Which method is used generally depends on physician preference. There have been no studies done to date that compare these two methods for needle insertion.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years and older
* Agreement to participate
* Patients with cirrhosis (confirmed by liver biopsy or clinically diagnosed) and ascites
* Patients presenting to UVA Digestive Health Clinic for a scheduled therapeutic paracentesis who do not have any contraindications to the procedure
* Ability to be reliably contacted by phone 24 hours following paracentesis

Exclusion Criteria:

* Prisoners
* Non-english speaking
* Paracentesis with less than 5 liters of ascitic fluid removed. (If this occurs, the specific subject encounter will be removed from the study but the subject may be included if at their next regularly scheduled paracentesis 5 liters or greater of ascitic fluid is removed.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2013-07; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Post procedural leaking at the needle insertion site | 24 hours

SECONDARY OUTCOMES:
Patient reported procedural pain | Immediately following paracentesis

CONTACTS AND LOCATIONS:
Overall Officials: Amy Rubin, MD, Principal Investigator — University of Virginia
Locations (1):
- University of Virginia, Charlottesville, Virginia, United States